CLINICAL TRIAL: NCT03937089
Title: Analysis of the Endocavitary Electrical Signal and Surface Electrocardiogram to Determine Relevant Features for an Accurate Prediction of Ablation Outcome for Patients in Persistent Atrial Fibrillation
Brief Title: Analysis of Endocavitary Electrical Signal and Surface Electrocardiogram to Predict Ablation Outcome in Persistent Atrial Fibrillation
Acronym: ASEPAF
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2018/ASEPAF-SELLAL/YB
Record Dates: First submitted 2019-04-08; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with persistent AF, who underwent a CA procedure in the Nancy hospital between January 2011 and April 2017, will be included in this retrospective study.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection from medical file

SUMMARY:
Background :

Despite recent progress in the management of patients with Atrial Fibrillation (AF), AF remains one of the main risk factor of stroke, heart failure and cardiovascular mortality in the world. AF is the most common cardiac arrhythmia, and its prevalence is expected to grow in the coming years.

Catheter ablation (CA) of AF can be successful in restoring and maintaining Sinus rhythm (SR) in patients with paroxysmal, and persistent AF. Haissaguerre et al. have shown that AF ablation of the heart by isolating the Pulmonary Vein is usually sufficient. However, when ablating persistent AF patients ablating pathological regions in the atria is also required. CA is still a challenging procedure, and reported success rate for persistent AF patients remains relatively low (around 60%). This procedure is associated with risks inherent to any invasive cardiac procedures.

A better identification of good responders would reduce the risks associated with ablation, especially for patients with low odds of favorable outcome, while also increasing the success rate of the procedure. It has been shown in the literature the long-term CA outcome can be predicted non-invasively by atrial fibrillatory wave (f-wave) amplitudes.

Hypothesis :

We assume that a morphological analysis of the f-waves on standard twelve ECG will allow for a better CA outcome prediction.

Objectives :

The aim of this study is to automatically analyse the morphology of the ECG signal before a CA procedure, extract relevant features for an accurate prediction of long-term CA outcome for patients in persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients for which clinical data, along with the ECG signals before and during the CA procedure are available,
* Patients who underwent a first ablation procedure for persistent AF

Exclusion Criteria:

* ECG data is not interpretable
* Patients who underwent a second or umpteenth ablation procedure for persistent AF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with persistent AF, who underwent a CA procedure in the Nancy hospital between January 2011 and April 2017, will be included in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of the f-waves on ECG | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France